CLINICAL TRIAL: NCT03009474
Title: Clinical Trial to Assess the Pharmacokinetic Characteristics of CJ-30060 in Healthy Male Subjects
Brief Title: Pharmacokinetics Study of CJ-30060 After Single Dose Administration in Health Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CJ_EXR_102
Record Dates: First submitted 2015-03-11; First posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Hypertension; Hyperlipidemias
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — Amlodipine, Valsartan Drug Combination; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CJ-30060 (Experimental): Amlodipine 5 mg/ Valsartan 160 mg/ Rosuvastatin 10 mg
  Interventions: Drug: Exforge tab 5/160mg, Crestor tab 10mg
- Exforge tab 5/160mg, Crestor tab 10mg (Active Comparator): Amlodipine 5 mg/ Valsartan 160 mg/ Rosuvastatin 10 mg
  Interventions: Drug: CJ-30060

INTERVENTIONS:
Drug: CJ-30060 — Fixed-dose combination drug containing Amlodipine 5 mg and Valsartan 160 mg and Rosuvastatin 10 mg
  Arms: Exforge tab 5/160mg, Crestor tab 10mg
Drug: Exforge tab 5/160mg, Crestor tab 10mg — Co-administration of Amlodipine 5 mg/ Valsartan 160 mg(combination drug) and Rosuvastatin 10 mg
  Arms: CJ-30060

SUMMARY:
To compare the pharmacokinetics and safety after a single dose administration of CJ-30060 and Exforge® 5/160mg, Crestor 10mg in healthy male volunteers.

DETAILED DESCRIPTION:
The purpose of this study is to compare the pharmacokinetics and safety after a single dose administration of CJ-30060 and Exforge® 5/160mg, Crestor 10mg in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male aged 20 to 45 years at the screening
* Subject who is over 50kg with BMI between 18 kg/m2 to 29 kg/m2 (inclusive)
* Subject who fully understood after being informed detailed description of clinical trial, written informed consent voluntarily to observe the precautions.

Exclusion Criteria:

* Subject who has a medical history of severe cardiovascular, respiratory, hepatobiliary, renal disease hematologic, gastrointestinal, endocrinological, immunologic, dermatosis or neuropsychologic disease.
* Subject who have symptoms, result from acute disease within 28days before first administration.
* Subject who have chronic persisting disease with clinical significance.
* Subject who fall under the criteria below in laboratory test.

  * AST/ALT > UNL (upper normal limit) x 2
  * Total bilirubin > UNL x 1.5
  * In case of renal failure that creatine clearance is less than 50mL/min according to Cockcroft-Gault
  * CPK > UNL x 2.5
* Subject who with low blood pressure with clinical significance at screening test.

(systolic blood pressure is less than 90 mmHg and diastolic blood pressure is less than 60 mmHg)

* Subject with any positive reaction in HBs Ag, anti-HCV Ab, anti-HIV Ab, VDRL tests.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of amlodipine, valsartan, rosuvastatin | Up to 144 hours post-dose

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of amlodipine, valsartan, rosuvastatin | Up to 144 hours post-dose
Time of maximum observed concentration (Tmax) of amlodipine, valsartan, rosuvastatin | Up to 144 hours post-dose
Half life (t1/2) of amlodipine, valsartan, rosuvastatin | Up to 144 hours post-dose
Oral clearance (CL/F) of amlodipine, valsartan, rosuvastatin | Up to 144 hours post-dose
Apparent volume of distribution (Vd/F) of amlodipine, valsartan, rosuvastatin | Up to 144 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Ji Young Park, PhD, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No